CLINICAL TRIAL: NCT07387562
Title: Mental Health Treatment in Caregivers of Psychiatric Patients: Application of Virtual Reality-Mediated Mindfulness
Brief Title: Virtual Reality-Based Mindfulness for Caregivers of Psychiatric Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Collaborators: Azienda Ospedaliero Universitaria Renato Dulbecco di Catanzaro (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 211/2025
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Caregivers; Caregivers Burnout
Keywords: caregivers; vr; virtual reality; mindfulness

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness and virtual reality (Experimental): To examine changes in psychological factors, the same psychometric tests will be administered to both groups before and after each intervention. This group participate in a 10-minute virtual reality-mediated mindfulness protocol.
  Interventions: Device: VR (VR-Control)
- Mindfulness and audio (Experimental): To examine changes in psychological factors, the same psychometric tests will be administered to both groups before and after each intervention. This group participate in a 10-minute immersive audio-mediated mindfulness protocol.
  Interventions: Device: Audio immersivo

INTERVENTIONS:
Device: VR (VR-Control) — Using the Meta Quest Pro headset, participants will participate in four virtual reality mindfulness exercises designed to improve relaxation and body awareness. Become's proprietary system (https://discoverbecome.com/) will be used for the sessions. The following is how the immersive "Augmented Wellbeing" sessions will be organized:
  1. observing the situation in "The Secret Garden";
  2. observing the "Sunset Beach" situation;
  3. observing the "Waterfall in the Meadow" situation; Reviewing the earlier sessions after viewing a scenario chosen by the participants to encourage self-determination and involvement.
  Arms: Mindfulness and virtual reality
Device: Audio immersivo — In order to improve body awareness and relaxation, participants will participate in four audio-only mindfulness sessions (immersive mindfulness audio). The same firm, BECOME, provides the audio track, which is the same as the one used in the VR immersive sessions. The number and length of sessions completed by participants will be identical to those of the experimental group, and the sessions will follow the same format:
  1. "The Secret Garden" immersive audio;
  2. "Sunset Beach" immersive audio;
  3. "Waterfall in the Meadow" immersive audio; Audio chosen by the participants to encourage participation and self-determination, followed by a recap of the earlier sessions.
  Arms: Mindfulness and audio

SUMMARY:
This clinical investigation aims to compare the mental health status of caregivers of psychiatric patients before and after virtual reality-based mindfulness. The study's primary objectives are to:

1. Does immersive audio-based mindfulness have a greater positive impact on psychological well-being than virtual reality-mediated mindfulness?
2. When compared to a single session, do four sessions lead to more improvements in psychological well-being? To assess the additional impact of virtual reality-mediated mindfulness, participants in the control group will receive mindfulness via immersive audio.

Those who voluntarily sign up for the study will participate in four sessions, one each week, on the same day and at the same time. Prior to and following the mindfulness intervention, self-administered psychometric assessment batteries will be completed.

While the control group will use ears to complete the mindfulness session using immersive audio, the experimental group will get a virtual reality-mediated mindfulness intervention. BECOME is the company that provides the audio and video content.

DETAILED DESCRIPTION:
In a sample of caregivers who visit the Department of Psychiatry at the "Renato Dulbecco" University Hospital in Catanzaro, the effects of the combined VR plus immersive audio treatment will be compared with the effects of immersive audio stimulation alone using a randomized controlled trial (RCT) design.

The main goal is to evaluate how much the experimental group's caregivers' mental health has improved both before and after therapy. The following self-report measures will be used for assessment: The World Health Organization Well-Being Index (WHO-5), the Zarit Burden Interview (ZBI), the Perceived Stress Scale (PSS-10), the Italian Mental Health Continuum-Short Form (MHC-SF), the Scale of Positive and Negative Experiences (SPANE), the Beck Depression Inventory-II (BDI-II), the State-Trait Anxiety Inventory (STAI), and the Pittsburgh Sleep Quality Index (PSQI).

Assessing variations in treatment effectiveness between the experimental and control groups is the secondary goal.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Being the primary caregiver of a psychiatric patient with a clinically confirmed diagnosis for at least 6 months.
* Willingness to participate for the entire duration of the study.
* Signed informed consent.

Exclusion Criteria:

* Active psychiatric diagnosis in the acute phase.
* Previous regular use of mindfulness techniques or other relaxation techniques at any point in life.
* Current use of psychotropic medications by the caregiver.
* Photosensitive epilepsy (due to VR headset use).
* Severe cognitive or sensory impairment.
* Binocular vision abnormalities.
* Hearing aids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) | From enrollment to the end of treatment at 4 weeks
Beck Depression Inventory (BDI-II) | From enrollment to the end of treatment at 4 weeks
Italian Mental Health Continuum - Short Form (MHC-SF) | From enrollment to the end of treatment at 4 weeks
Perceived Stress Scale (PSS-10) | From enrollment to the end of treatment at 4 weeks
WHO-5 | From enrollment to the end of treatment at 4 weeks
Mindful Attention Awareness Scale (MAAS) | From enrollment to the end of treatment at 4 weeks
Zarit Burden Interview (ZBI) | From enrollment to the end of treatment at 4 weeks
Scale of Positive and Negative Experiences (SPANE) | From enrollment to the end of treatment at 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- AOU "Renato Dulbecco", Catanzaro, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: No